CLINICAL TRIAL: NCT01457651
Title: Comparison of Different Types of Postoperative Pulmonary Recruitment and Predicting Its Efficacy Following Off-pump Coronary Artery Bypass Grafting
Brief Title: Comparison of Four Different Recruitment Maneuvers in Patients After Coronary Surgery
Acronym: RECR-CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Collaborators: Regional hospital of Arkhangelsk (Unknown)
Responsible Party: Principal Investigator, Vsevolod V. Kuzkov, Associate Professor, MD, PhD, Northern State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECR-CABG-2010
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Hypoxemia; Recruitment
Keywords: Recruitment; Coronary artery bypass grafting; Postoperative period
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Recruitment 40x40 (Active Comparator): The group where recruitment is performed by increase in airway pressure up to 40 cm H2O for 40 seconds
  Interventions: Procedure: Alveolar recruitment
- Recruitment PEAK40 (Active Comparator): Increase in peak airway pressure up to 40 cm H2O during tidal ventilation
  Interventions: Procedure: Alveolar recruitment
- Recruitment 15x300 (Active Comparator): Recruitment by increase in airway PEEP up to 15 cm H2O for 300 sec
  Interventions: Procedure: Alveolar recruitment
- No recruitment (Active Comparator): No recruitment is performed: standard respiratory support.
  Interventions: Procedure: Alveolar recruitment

INTERVENTIONS:
Procedure: Alveolar recruitment — Four approaches:
  1. CPAP 40 cm H2O
  2. Peak pressure 40 cm H2O
  3. PEEP 15 cm H2O for 300 sec
  4. no intervention (controls)
  Other Names: CPAP40; PEAK40; PEEP15; CONTROLS

SUMMARY:
The risk of respiratory failure after cardiac surgery is high, and it may result in many complications. The maneuver of alveolar recruitment may improve the oxygen transport in the human organism. The investigators compare three different types of alveolar recruitment in patient after cardiac surgery, to reveal which one is better.

DETAILED DESCRIPTION:
The study compares three different approaches to alveolar recruitment maneuvers in the immediate postoperative period after off-pump coronary bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75
* Off-pump coronary artery bypass grafting
* Possibility to discontinue respiratory support in the first day after intervention

Exclusion Criteria:

* Signs of ARDS
* COPD in decompensation phase
* Requirement for inotropic support(epinephrine >0,1 mcg/kg/hr)
* Bronchiectases
* Pregnancy
* Morbid obesity
* Aortic aneurism
* AMI in previous month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Respiratory support | 24 hrs
  The duration of the postoperative respiratory support

SECONDARY OUTCOMES:
The incidence of postoperative atelectasis | 24 hrs
  Incidence of atelectases during 24 hrs
Incidence of reintubation | 24 Hrs
Oxygenation | 12 hrs after extubation
  Changes in PaO2/FiO2 ratio
Length of ICU and hospital stay | 28 Days
  Length of ICU and hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y. Kirov, MD, PhD, Study Director — Northern State Medical University
Locations (1):
- City hospital # 1, Arkhangelsk, Arkhangelskaya oblast, Russia